CLINICAL TRIAL: NCT00399425
Title: Triple-Blind Clinical Trial With Placebo Control to Evaluate the Efficacy of a Heparin of Low Molecular Weight (Bemiparin) for Treating Slow-Responding Ulcers in Diabetic Foot in Primary Care
Brief Title: Efficacy of a Low-Molecular-Weight Heparin (Bemiparin) in the Treatment of Chronic Foot Ulcers in Diabetic Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Spanish National Health System (Other)
Collaborators: Carlos III Health Institute (Other Government); Rovi Pharmaceuticals Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APM/00/PD1; AEM 01-0167
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Foot Ulcer, Diabetic; Diabetic Angiopathies
Keywords: Heparin, Low-Molecular-Weight; Bemiparin; Foot Ulcer, Diabetic; Diabetic Angiopathies; Primary Health Care
MeSH Terms: conditions — Diabetic Foot; Diabetic Angiopathies | interventions — bemiparin; Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: bemiparin (low molecular weight heparin)

SUMMARY:
To assess the efficacy of bemiparin (low molecular weight heparin) for 3 months in the treatment of chronic foot ulcers in diabetic patients.

DETAILED DESCRIPTION:
The involvement of microcirculation in diabetes microangiopathy may be the cause of ulceration and severe incapacitation. Torpid ulcers of the lower limbs affect up to 15% of diabetic patients at some moment of their lifetime; about one-third of patients developing ulcers will never achieve their definitive cure, and half of them will die within three years .

Heparins, besides their well known antithrombotic effects, have been shown to stimulate both the synthesis of heparan sulphate -a potent endogenous anticoagulant- in endothelial cell cultures and the proliferation of fibroblasts taken from diabetic ulcers .

After noticing the highly positive evolution of chronic ulcers in six diabetic patients who had received LMWHs in their homes for the prophylaxis of deep vein thrombosis , and considering the excellent safety record of these drugs, we decided to explore the effects of LMWHs on the evolution of diabetic foot ulcers and the quality of life of diabetic patients seen in our primary care practices.

Comparison: bemiparin vs placebo

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* type I or II diabetes mellitus diagnosed (ADA 1998) for more than 3 years;
* presence of at least one cutaneous ulcer distal to the knee, not involving deep tissues (stages I and II of Wagner's classification ) and existing for at least three months;
* giving their written informed consent.

Exclusion Criteria:

* hypersensibility to heparin or pig derivatives
* body weight lower than 35 kg
* presence of clinical signs of infection that did not resolve in spite of oral antibiotics;
* anticoagulant therapy;
* severe impairment of renal or hepatic function;
* bleeding disorder;
* active peptic ulcer;
* arterial hypertension with poor control;
* pregnancy or lactation;
* terminal illness or a prognosis of survival under three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2001-06; Study Completion 2004-04

PRIMARY OUTCOMES:
Ulcer area
Stage in Wagner's classification

SECONDARY OUTCOMES:
Adverse effects
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rullan, MD, Principal Investigator — Primary health care of Mallorca. Ibsalut.

REFERENCES:
- [Background] Rullan M, Cerda L, Frontera G, Llobera J, Masmiquel L, Olea JL. [Triple-blind clinical trial with placebo control to evaluate the efficacy of a heparin of low molecular weight (bemiparin) for treating slow-responding ulcers in diabetic foot in primary care]. Aten Primaria. 2003 May 15;31(8):539-44. doi: 10.1016/s0212-6567(03)70729-x. Spanish. PMID 12765594